CLINICAL TRIAL: NCT04617002
Title: Intermediate-size Expanded Access to ONC201 for Patients With H3 K27M-mutant and/or Midline Gliomas
Status: Approved for marketing | Type: Expanded Access
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ONC028
Record Dates: First submitted 2020-10-29; First posted 2020-11-05 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Glioma; H3 K27M
MeSH Terms: conditions — Glioma | interventions — TIC10 compound

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: ONC201 (dordaviprone) — ONC201 (dordaviprone) is a ClpP agonist and DRD2 antagonist.

SUMMARY:
This is an intermediate-size expanded access protocol to provide ONC201 (dordaviprone) to patients with H3 K27M-mutant and/or midline gliomas who cannot access ONC201 (dordaviprone) through clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Patient meets one or more of the criteria below:

   Arm A - Closed to further enrollment.

   Arm B - Diffuse intrinsic pontine glioma (DIPG) defined as tumors with a pontine epicenter and diffuse involvement of the pons (at the discretion of the Medical Monitor, the site may be requested to provide the most recent imaging report(s) to confirm diagnosis). H3 K27M status does not have to be known or positive for this arm.

   Arm C -
   1. Patients with primary spinal glioma that is positive for the H3 K27M mutation (performed in a laboratory with Clinical Laboratory Improvement Amendments [CLIA] or equivalent certification). Primary spinal glioma must be documented in radiology reporting.

      OR
   2. Patients with diffuse glioma that is positive for the H3 K27M mutation (performed in a laboratory with CLIA or equivalent certification) AND radiographic evidence of leptomeningeal disease. Leptomeningeal disease must be documented in radiology reporting.

   Arm D - Closed to further enrollment.

   Arm E - Patients with H3 K27M-mutant glioma or a midline glioma of unknown H3 K27M mutational status who received ONC201 and/or ONC206 from an alternative (non-Chimerix) source prior to 31 December 2023, as evidenced by supporting documentation (e.g., medical records, pharmacy receipts, etc.). Other supporting documentation may be confirmed by the medical monitor. Detection of H3 K27M mutation should be performed in a CLIA-certified or equivalent laboratory.

   Arm F - Patients with H3 K27M-mutant diffuse glioma who have progressed during or after completion of frontline radiotherapy. Detection of H3 K27M mutation should be performed in a CLIA-certified or equivalent laboratory. Enrollment in this arm will be individually evaluated by the Sponsor and requires at least 3 days for review.
2. Disease status:

   Arm B - Patient is not required to have radiographic or clinical evidence of progressive disease.

   Arm C - Patient must have progressive disease as defined by Response Assessment in Neuro-Oncology (RANO) criteria or have documented recurrent glioma on diagnostic biopsy.

   Arm E - Not applicable.

   Arm F - Patient must have progressive disease as defined by RANO criteria or have documented recurrent glioma on diagnostic biopsy.
3. Prior radiotherapy:

   Arm B - Patient must be at least 14 days from completion of radiotherapy.

   Arm C - Patient must be at least 30 days from completion of frontline radiotherapy and at least 14 days from reirradiation if applicable.

   Arm E - Not applicable.

   Arm F - Patient must be at least 30 days from completion of frontline radiotherapy and at least 14 days from reirradiation if applicable.
4. (Not applicable; criterion removed in Version 5).
5. Patients must weigh at least 10 kg.
6. Washouts:

   Arms B, C, and F - From the projected start of scheduled study treatment, the following time periods must have elapsed from prior anti-cancer treatments: 5 half-lives from any investigational agent, 4 weeks from cytotoxic therapy (except 23 days for temozolomide and 6 weeks from nitrosoureas), 6 weeks from anti-cancer antibodies (no washout required for bevacizumab), 4 weeks (or 5 half-lives, whichever is shorter) from other anti-tumor therapies including CAR-T and other cellular therapies/immunotherapies, and 1 week from devices used to treat cancer.

   Arm E - No washouts are required for ONC201 and ONC206. All other anti-cancer agents need to be discontinued prior to enrollment with the exception of bevacizumab.
7. Magnetic resonance imaging (MRI) of patient's glioma obtained within 28 days prior to start of ONC201 for Arms B, C, and F.

   Arm E: MRI obtained within 8 weeks prior to enrollment.
8. Adequate organ and marrow function as defined below:

   1. Absolute neutrophil count ≥1,000/mm3 without growth factor use ≤7 days prior to treatment (Cycle 1 Day 1 [C1D1])
   2. Hemoglobin ≥8.0 mg/dL without red blood cell transfusion ≤3 days prior to C1D1
   3. Total serum bilirubin ≤1.5 X upper limit of normal (ULN) (participants with Gilbert's syndrome may be included with total bilirubin > 1.5 × ULN if direct bilirubin is ≤ 1.5 × ULN)
   4. AST (SGOT)/ALT (SGPT) ≤2.5 X ULN; ≤5 X ULN if there is liver involvement secondary to tumor
   5. Serum creatinine ≤1.5 X ULN (OR creatinine clearance ≥60 mL/min/1.73 m2) Arm E: Patients with organ and marrow function laboratory values outside the defined criteria must be approved by the medical monitor.
9. Female patients of childbearing potential must agree to use an effective contraception method while taking ONC201 and for at least 90 days after the last dose of ONC201 and must have a negative pregnancy test prior to starting ONC201. Male patients must be surgically sterile (i.e., >3 months post-vasectomy) or must agree to use an effective contraception method while taking ONC201 and for at least 90 days after the last dose of ONC201. Determination of effective contraception methods will be based on the judgment of the Investigator.
10. Ability to understand a written informed consent document, and the willingness to sign it. At the discretion of the Investigator, a Legally Authorized Representative (LAR) may consent on behalf of a patient who is unable to provide informed consent themselves. Assent will be obtained, as appropriate, based on the patient's age.

Exclusion Criteria:

1. Qualifies for participation in an ongoing ONC201 or ONC206 clinical trial.
2. Arms B, C, and F: Previous or current enrollment in an ONC201 or ONC206 clinical study (including open-label and blinded studies) or expanded access protocol or previous exposure to ONC201 from any source for the treatment of CNS tumor.

   Arm E: Previous or current enrollment in an ONC201 clinical study (including open label and blinded studies) or expanded access protocol for the treatment of CNS tumor.
3. Current or planned participation in a study of an investigational agent (including ONC206) or using an investigational device.
4. (Not applicable; criterion removed in Version 4).
5. Any known systemic infection that, in the opinion of the Investigator, could compromise the safety of the patient while taking ONC201.
6. Prolongation of QT/QTcF interval (QTc interval >480 milliseconds) using Fridericia's QT correction formula on two electrocardiograms (ECGs) separated by at least 2 days.
7. A history of Torsades de pointes or heart failure, hypokalemia, or family history of prolonged QT Syndrome.
8. Concomitant use of medication(s) known to prolong the QT/QTc interval.

Min Age: 0 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - BMDACC at Banner University Medical Center Phoenix, Phoenix, Arizona
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Rady Children's Hospital, San Diego, California
  - Providence Saint John's Health Center, Santa Monica, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Miami Cancer Institute, Miami, Florida
  - University Cancer & Blood Center, Athens, Georgia
  - Kapi'olani Medical Center for Women and Children, Honolulu, Hawaii
  - Lurie Children's Hospital, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center - Adults Only, Omaha, Nebraska
  - Overlook Medical Center/ Atlantic Health System, Summit, New Jersey
  - Albany Medical Center, Albany, New York
  - New York University Langone - Active, Enrolling, New York, New York
  - University of Rochester, Rochester, New York
  - Providence Neurological Specialties Clinic, Portland, Oregon
  - University of Texas Southwestern, Dallas, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia